CLINICAL TRIAL: NCT01763931
Title: Digoxin as a Novel Inhibitor of Global Hypoxia Inducible Factor-1α (HIF-1α) Expression & Downstream Targets in Breast Cancer: DIG-HIF-1 Pharmacodynamic Trial
Brief Title: DIG-HIF-1 Pharmacodynamic Trial in Newly Diagnosed Operable Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: J1232; A-17427 (Other: Department of Defense (DoD)); NA_00072292 (Other: JHMIRB)
Record Dates: First submitted 2013-01-07; First posted 2013-01-09 (Estimated); Results first posted 2020-01-31 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Breast Cancer
Keywords: Digoxin
MeSH Terms: conditions — Breast Neoplasms | interventions — Digoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Digoxin (Experimental): Digoxin administration for 2 weeks prior to surgery.
  Interventions: Drug: Digoxin
- No drug administration prior to surgery (No Intervention): Group of participants who will not receive digoxin; however, tissue will be collected at time of definitive breast surgery.

INTERVENTIONS:
Drug: Digoxin — Digoxin once daily for 2 weeks prior to definitive breast surgery.
  Arms: Digoxin

SUMMARY:
The purpose of this study is to learn what effects digoxin (DIG) may have on human breast cancer tissue.

DETAILED DESCRIPTION:
Breast cancer cells grow in a low oxygen environment called hypoxia. The body normally controls the amount of oxygen in cells with what is known as Hypoxia-inducible factor (HIF)-1. HIF-1 helps cancer cells grow in low oxygen environments; therefore, if this function can be blocked, it may make it harder for breast cancer cells to grow. Digoxin is a drug that has been shown to block HIF-1 in lab studies. The investigators want to learn if it blocks HIF-1 in human breast cancer tissue. This will be done by comparing the tumor tissue from the original diagnostic biopsy to tissue that is taken at the time of surgery. The investigators will also be comparing tumor tissue of patients who are not randomized to take digoxin.

ELIGIBILITY:
Inclusion Criteria:

* Female sex
* 18-70 years of age at time of consent.
* Histologically confirmed infiltrating carcinoma of the breast (Stage I-III)
* Unresected disease that meets scheduled to undergo definitive surgery; tumor size ≥ 1cm; grade 2 or 3 tumor or Ki-67 proliferation index of ≥ 10%; and, any estrogen receptor (ER), progesterone receptor (PR) or human epidermal growth factor receptor 2 (HER2) status
* Patients must not have received any prior treatment of any kind to treat the current breast cancer.
* Prior use of hormone contraceptives and replacement therapy is allowed, but must have been discontinued at least 30 days prior to the diagnostic biopsy.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 (Karnofsky 80%-100%)
* Patients must have normal organ and marrow function: absolute neutrophil count (ANC) ≥ 1,500/mm3; platelet count ≥ 100,000/mm3; bilirubin (total) less than or equal to the upper limit of normal; creatinine ≤ 1.5 times the upper limit of normal with creatinine clearance ≥ 50 mL/min using the Modified Cockcroft-Gault method; and, all of the following within normal limits: thyroid stimulating hormone (TSH), magnesium, potassium, sodium, calcium.
* Heart rate > 60 beats/minute and < 100 beats/minute (clinical exam).
* Not pregnant or nursing
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Current use of any investigational agents
* Radiological evidence of metastatic disease
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to digoxin
* Concomitant use of these drugs at baseline and for the duration of digoxin administration (if randomized to receive it): the calcium channel blockers diltiazem or verapamil; cardiac arrhythmic agents (such as quinidine, amiodarone); indomethacin (Indocin); alprazolam (Xanax); diuretics (such as furosemide, spironolactone, itraconazole); beta-blockers (such as atenolol, metoprolol); calcium carbonate antacids (e.g., Maalox, Tums, Rolaids); proton pump inhibitors; antidiarrheal adsorbents (kaolin and pectin); antibiotics; other P450 inducer/inhibitors. Note: Patients already receiving digoxin are also excluded.
* Presence of any of the following on electrocardiogram (ECG): atrial arrhythmias, including atrial fibrillation and flutter; AV block; heart rate < 60 beats/minute and > 100 beats/minute; ventricular Fibrillation; ventricular tachycardia; premature ventricular contractions; Wolff-Parkinson-White syndrome. Note: Any questions on cardiac eligibility should be reviewed by the Study Cardiologist for approval in advance of enrollment.
* History of any of the following, unless approval is given by the Protocol Chair: heart disease, including acute myocardial infarction; cardiac arrhythmias, including sick sinus syndrome; pulmonary disease with a known forced expiratory volume (FEV) of <1.5 or on oxygen; gastrointestinal disease, surgery or malabsorption that could potentially impact the absorption of the study drug; patients requiring the use of a feeding tube; inability to swallow tablets
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that will limit compliance with study requirements
* Any medical condition which in the opinion of the investigator puts the patient at risk of potentially serious complications while on this therapy

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-01; Primary Completion 2016-04-01 (Actual); Study Completion 2016-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vered Stearns, M.D., Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Kimmel Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Digoxin | No Drug Administration Prior to Surgery
Started | 2 | 4
Completed | 2 | 3
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Digoxin | No Drug Administration Prior to Surgery | Total
Number analyzed (Participants) | 2 | 4 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 4 | 5
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Full Range); unit: years] | 65 [63 to 66] | 44 [27 to 62] | 51 [27 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 2 | 3 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race - White | 2 | 1 | 3
  Race - Black | 0 | 1 | 1
  Race - Other | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in HIF-1α Protein Expression
Description: To assess whether two weeks of daily oral digoxin therapy, as compared to no study drug, reduces the expression of Hypoxia-inducible factor (HIF)-1α protein, measured by immunohistochemistry (IHC), in surgically resected breast cancer tissue obtained from women undergoing lumpectomy or mastectomy for invasive breast cancer.
Time Frame: Baseline (biopsy prior to surgery) and at the end of 2 weeks digoxin treatment
Population: Not enough tissue samples were collected to be analyzed and so no data was generated for this outcome measure.
Arm/Group | Digoxin | No Drug Administration Prior to Surgery
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Number of Participants With Adverse Events With Digoxin Treatment
Description: To assess safety and tolerability of two weeks of digoxin therapy in the pre-surgical setting graded according to Common Terminology Criteria for Adverse Events (CTCAE), version 4.
Time Frame: 2 weeks
Population: Adverse events with digoxin is not applicable to the group "no drug administration prior to surgery"
Measure: Count of Participants; unit: Participants
Arm/Group | Digoxin | No Drug Administration Prior to Surgery
Number analyzed (Participants) | 2 | 0
Participants | 2 | 0

ADVERSE EVENTS:
Arm/Group | Digoxin | No Drug Administration Prior to Surgery
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/4
Other Adverse Events (participants affected / at risk) | 2/2 | 0/4
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Digoxin (N=2) | No Drug Administration Prior to Surgery (N=4)
Hip Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Grade 1, unrelated
Ear Pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) — Grade 1, unrelated
Incisional pain (Surgical and medical procedures) | 2 (2) | 0 (0) — Maximum grade 2, unrelated to study drug
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) — Grade 1, possibly related
Increased urine output (Renal and urinary disorders) | 1 (1) | 0 (0) — Grade 1, possibly related
Knee pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Grade 1, unrelated
Neck spasms/pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Grade 2, unrelated
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) — Grade 2, unrelated

LIMITATIONS AND CAVEATS:
The pre-operative setting was challenging for accrual and we did not meet our accrual goals. Therefore, the study was closed to accrual early. Only 6 out of 64 planned participants were enrolled, therefore there was not enough data to analyze.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No